CLINICAL TRIAL: NCT01421368
Title: Assessing the Effect of Contraception and the Menstrual Cycle on Pharmacokinetics, Pharmacodynamics, and Vaginal Safety in Tenofovir Vaginal Gel Users
Brief Title: Contraception and Menstrual Cycle Effect on Pharmacokinetics, Pharmacodynamics and Safety in Tenofovir Vaginal Gel Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A10-114
Record Dates: First submitted 2011-08-09; First posted 2011-08-22 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Tenofovir; Vaginal Creams, Foams, and Jellies; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMPA and tenofovir 1% gel (Experimental)
  Interventions: Drug: Tenofovir 1% vaginal gel; Drug: Depo-medroxyprogesterone acetate (DMPA)
- Oral contraceptive and tenofovir 1% gel (Experimental)
  Interventions: Drug: Tenofovir 1% vaginal gel; Drug: Oral contraceptive: LNG 150 mcg and EE 30 mcg

INTERVENTIONS:
Drug: Tenofovir 1% vaginal gel — Tenofovir 1% gel is supplied as a clear, transparent, viscous gel packaged in pre-filled single use applicators. Each applicator contains 4.0 mL of tenofovir gel (equal to 4.4 gm) at a concentration of 1% (weight for weight) formulated in purified water with edetate disodium, citric acid, glycerin, methylparaben, propylparaben and hydroxyethylcellulose, and is pH adjusted to 4-5
Drug: Depo-medroxyprogesterone acetate (DMPA) — DMPA is an intramuscular injectable contraceptive containing 150 mg of medroxyprogesterone acetate. It is FDA approved for 12 weeks of use per injection.
  Other Names: Depo-Provera
  Arms: DMPA and tenofovir 1% gel
Drug: Oral contraceptive: LNG 150 mcg and EE 30 mcg — Each pill contains LNG 150 mcg (the active levorotatory enantiomer of norgestrel) and EE 30 mcg. Each pack contains 21 active pills and 7 placebo pills
  Arms: Oral contraceptive and tenofovir 1% gel

SUMMARY:
The purpose of the study is to examine the effects of two contraceptive methods and the menstrual cycle on the pharmacokinetics, pharmacodynamics of tenofovir 1% gel and the effect of the contraceptive methods on markers of mucosal safety.

DETAILED DESCRIPTION:
Each woman will be seen in 6 visits and will be contacted by two scheduled follow-up telephone calls/visits. Volunteers will be consented at Visit 1 and undergo procedures to assess whether they are eligible to continue in the study. At Visit 2 (cycle days 20-25), after it has been confirmed that the participant meets all of the inclusion criteria and none of the exclusion criteria, genital samples will be taken and she will be given 2 applicators of tenofovir 1% gel to insert two hours apart. She will be instructed to return for Visit 3, approximately 3 or 11 hours after insertion of the second gel, as determined by randomization. The participant will retain this sampling assignment throughout the study.

At Visit 3 (cycle days 20-25), blood and genital samples will be collected. The participant will again be given 2 applicators of tenofovir 1% gel to insert two hours apart. She will be instructed to return approximately 3 or 11 hours after insertion of the second gel for Visit 4 (cycle days 5-10) and blood and genital samples will be taken. The participant will then start the contraceptive method that she has chosen from the two methods being evaluated in the study.

Each participant will be contacted about 4-5 weeks after Visit 4 to confirm the next visit date (Visit 5).

Visit 5 will take place about 6 weeks after starting contraception and will not have an associated gel use. Follow-up genital samples will be collected at Visit 5. The participant will be given 2 applicators of tenofovir 1% gel to insert two hours apart prior to Visit 6.

Visit 6 will take place about 10 weeks after starting contraception. Follow-up blood and genital samples will be collected approximately 3 or 11 hours after insertion of the second gel.

Each participant also will have a follow-up call or visit approximately 1-2 weeks after Visit 6 to confirm that there have been no adverse experiences. If necessary, she may be seen in an unscheduled visit for follow-up. She will then be exited from the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to use OCs or DMPA
* General good health (by volunteer history and investigator assessment) without any clinically significant systemic disease
* Currently having regular menstrual cycles of 25 to 35 days by volunteer report
* History of Pap smears and follow-up consistent with American Congress of Obstetricians and Gynecologists (ACOG) practice bulletin #99 or #109 or willing to undergo a Pap smear at Visit 1
* Willing to follow protocol requirements including abstinence, use of study condoms, and prohibited use of intravaginal products
* Willing to follow post-biopsy restrictions for at least 5 days following genital biopsies
* Meets one of the following criteria:

  1. Sexually abstinent and planning to remain abstinent for the duration of the study.
  2. In a mutually monogamous relationship for at least the last 4 months with a male partner who is at least 18 years of age, willing to use condoms, and has no known HIV infection or risks for sexually transmitted infections (STIs)
  3. In a mutually monogamous same-sex relationship for at least the last 4 months with a partner who is at least 18 years of age and has no known HIV infection or risks for STIs
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy genital tract sample collection
* Negative urine pregnancy test
* Willing to give voluntary consent, sign an informed consent form and comply with study procedures, as required by the protocol

Exclusion Criteria:

* History of hysterectomy
* Currently pregnant or within 2 calendar months from the last pregnancy outcome. (Note: If recently pregnant must have had at least 2 spontaneous menses since pregnancy outcome.)
* Use of any hormonal contraceptive method in the last 30 days (oral, transdermal, transvaginal, implant, or hormonal intrauterine contraceptive device)
* Injection of DMPA in the last 6 months
* Protection from pregnancy by presence of a copper IUD
* Currently breastfeeding or having breastfed an infant in the last 2 months, or planning to breastfeed during the course of the study
* History of sensitivity/allergy to any component of the study product, or topical anesthetic, or allergy to both silver nitrate and Monsel's solution
* Diagnosed with or treated for any STI or pelvic inflammatory disease in the last 6 months. (Note: Women with a history of genital herpes or condylomata who have been asymptomatic for at least 6 months may be considered for eligibility.)
* Positive test for Trichomonas vaginalis, Neisseria gonorrhoeae or Chlamydia trachomatis
* Symptomatic vulvovaginal candidiasis, Nugent score greater than or equal to 7 at screening or bacterial vaginosis (BV) at Visit 2, or urinary tract infection (UTI)
* Deep epithelial genital findings such as abrasions, ulcerations, or lacerations, or vesicles suspicious for STIs
* Positive test for HIV
* Positive test for Hepatitis B surface antigen (HBsAg)
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy
* Chronic or acute vulvar or vaginal symptoms (e.g., pain, irritation, or spotting)
* Contraindications to the chosen contraceptive method
* Known current drug or alcohol abuse which could impact study compliance
* Grade 1 or higher laboratory abnormality, per the August 2009 update of the DAIDS Table for Grading the Severity of Adverse Events
* Participation in any other investigational trial (device, drug, or vaginal trial) in the last 30 days or planned participation in any other investigational trial during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix in the last 14 days
* Abnormal finding on laboratory or physical examination or a social or medical condition which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, antifungals, antivirals or antiretrovirals

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Effect of oral contraceptives and DMPA on tenofovir PK, PD, and safety by comparing the following endpoints before initiation of contraceptive method and 10 weeks after initiation of contraceptive method | 3 and 11 hours after insertion of 2 doses of study gel
  * composite of pharmacokinetics for TFV in plasma, vaginal aspirate & genital tissue
  * composite of pharmacokinetics for TFV-DP in PBMCs, endocervical cells & genital tissue
  * rates of HIV-1 infection in an explant challenge assay (one site only)
  * immune cell activation & mucosal histology in genital tissue
  * genitourinary AEs

SECONDARY OUTCOMES:
Effect of the menstrual cycle of the tenofovir PK, PD, and safety by comparing the following endpoints 3 and 1 hours after insertion of 2 doses of study gel, in the follicular and luteal phases before initiating contraception | 3 and 11 hours after insertion of 2 doses of study gel
  * composite of pharmacokinetics for TFV in plasma, vaginal aspirate & genital tissue
  * composite of pharmacokinetics for TFV-DP in PBMCs, endocervical cells & genital tissue
  * rates of HIV-1 infection in an explant challenge assay (one site only)
  * immune cell activation & mucosal histology in genital tissue
  * genitourinary AEs
To assess the effect of oral contraceptives and DMPA on markers of mucosal immunity by comparing the following endpoints (in the absence of tenofovir) before initiation of contraceptive method and 10 weeks after initiation of contraceptive method | Before (baseline) and 10 weeks after contraceptive method start
  * soluble immune markers in the CVL supernatant
  * anti-HIV and anti-HSV in CVL
  * immune cell characterization in the CVL cell pellet
  * immune cell activation and mucosal histology in genital tissue
  * rates of HIV-1 infection in an explant challenge assay (one site only)
  * vaginal microflora
  * genitourinary AEs

CONTACTS AND LOCATIONS:
Overall Officials: Christine K. Mauck, M.D., Study Director — CONRAD
Locations (3):
- United States (2):
  - University of Pittsburgh School of Medicine, Center for Family Planning Research, Pittsburgh, Pennsylvania
  - Easter Virginia Medical School, Norfolk, Virginia
- Profamilia, Santo Domingo, Dominican Republic

REFERENCES:
- [Derived] Zalenskaya IA, Chandra N, Yousefieh N, Fang X, Adedipe OE, Jackson SS, Anderson SM, Mauck CK, Schwartz JL, Thurman AR, Doncel GF. Use of contraceptive depot medroxyprogesterone acetate is associated with impaired cervicovaginal mucosal integrity. J Clin Invest. 2018 Oct 1;128(10):4622-4638. doi: 10.1172/JCI120583. Epub 2018 Sep 17. PMID 30222141